CLINICAL TRIAL: NCT05847816
Title: The Effects of Three Different Techniques During Peripheral Intravenous Cannulation (PIVC) Administered in Vein Visibility, Pain and Comfort in Cancer Patients Receiving Palliative Care
Brief Title: The Effects of Three Different Techniques During PIVC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Hulya Yilmaz, PhD, Principal Investigator, PhD, Msc, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 28/09/2022 - 713/693
Record Dates: First submitted 2023-04-03; First posted 2023-05-08 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Pain; Arm; Visual Aura; Infrared; Rays, Injury
Keywords: near-infrared light; peripheral intravenous cannulation; pain; arm comfort
MeSH Terms: conditions — Pain; Epilepsy, Partial, Sensory; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized controlled experimental study.
Masking Description: The intervention and measurements will carried out by the TY (for hand manipulation standard) and the patients will discovered their own groups when intervention will applied to them. Because of the nature of the intervention, blinding will not be performed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group: infrared vascular imaging (Experimental): The patient's vital signs, skin color and skin turgor will be evaluated and recorded in the peripheral intravenous chemotherapy application registration form. After the tourniquet is attached, the stopwatch will be started and the catheter intervention process will be started when the vein visibility reaches the level where the nurse can insert the catheter. The stopwatch will be terminated at the stage of advancing the branule into the vein and fixing it with a plaster. If the catheterization application is successful or unsuccessful in the first attempt, it will be recorded. The pain and arm comfort levels in the form will be evaluated on a scale ranging from 0 to 10, with 0: none, 10: many, before and after the application (at the 5th, 30th, and 60th minutes).
  Interventions: Other: Experimental group: infrared vascular imaging
- Experimental group: isometric hand exercise (Experimental): The patients to be included in this group will have applied isometric hand squeeze exercise, which lasted for twenty minutes a day, five days a week, before the PIVK procedure. On the fifth day, the patient's vital signs, skin color and skin turgor will be evaluated and recorded in the peripheral intravenous chemotherapy application registration form. Patients will be told how to use the stress ball 5 minutes before and during the PIVK procedure before the procedure. Patients will be taught to count from one to three and tighten and loosen the stress ball once, and they will be told to continue squeezing and loosening the stress ball in this way until the procedure is over. Focus their attention on the stress ball during the procedure.
  Interventions: Other: Experimental group: infrared vascular imaging
- Control group: no intervention (No Intervention): The patient's vital signs, skin color and skin turgor will be evaluated and recorded in the peripheral intravenous chemotherapy application registration form. After the tourniquet is attached, the stop watch will be started and the catheter intervention process will be started when the vein visibility reaches the level where the nurse can insert the catheter. If the PIVC application is successful or unsuccessful in the first attempt, it will be recorded. PIC success will be evaluated according to whether the branule is placed in the vein. The pain and arm comfort levels in the form will be evaluated on a scale ranging from 0 to 10, with 0: none, 10: many, before and after the application (at the 5th, 30th, and 60th minutes).

INTERVENTIONS:
Other: Experimental group: infrared vascular imaging — Experimental group - infrared vascular imaging;Before PIVC, infrared light will be directed to the vein area and the procedure will be started after vein visibility is achieved.
  Experimental group - isometric hand exercise; Stress balls will be given to patients 10 minutes before the PIVC procedure and they will be asked to perform hand-clamping exercises with both hands. Processing will then begin.
  Other Names: Experimental group: isometric hand exercise
  Arms: Experimental group: infrared vascular imaging; Experimental group: isometric hand exercise

SUMMARY:
Purpose: This study will conducted to the effect of three different techniques used during peripheral intravenous cannulation (PIVC) application on vein visibility, pain and comfort in cancer patients receiving palliative care.

Design: This is a prospective, randomized controlled experimental study. Methods: The population of the research will be cancer patients who applied to Ege University Medical Faculty Hospital Oncology unit between April 2023 and November 2024. The number of applications due to palliative care and cancer treatment in the clinic in 2021 is 352 patients. For this reason, direct sample selection was not made in the study, and the sample calculation was made according to the number of patients registered in the unit and the results of previous research (Chiao et al., 2013; Aulagnier et al., 2014). Calculations were made using the "G.Power-3.17" program with 95% confidence, an effect size of 0.4, and a statistical test power of at least 80%. Accordingly, it was aimed to reach 120 patients, including at least 40 in each group. In the study, randomization will be made according to vein visibility.

DETAILED DESCRIPTION:
Purpose: This study will conducted to the effect of three different techniques used during peripheral intravenous cannulation (PIVC) application on vein visibility, pain and comfort in cancer patients receiving palliative care. We will implement of the study during the insert on PIVC; the vascular imaging device group; isometric hand exercise group and control group.

Design: This is a prospective, randomized controlled experimental study.

Methods: Implementation of the study in the control group: The patient's vital signs, skin color and skin turgor will be evaluated and recorded in the peripheral intravenous chemotherapy application registration form. Since it is stated in the literature that the placement of the PIVK in the arm that is not actively used is important in preventing complications, PIVK will be placed in the arm that the patient does not actively use in groups (Ingram and Lavery, 2005; INS, 2011). After the tourniquet is attached, the stopwatch will be started and the catheter intervention process will be started when the vein visibility reaches the level where the nurse can insert the catheter. The stopwatch will be terminated at the stage of advancing the branule into the vein and fixing it with a plaster. If the catheterization application is successful or unsuccessful in the first attempt, it will be recorded. PIC success will be evaluated according to whether the branule is placed in the vein. Successful catheter insertion will be considered as blood coming into the chamber of the catheter. If the vein cannot be entered or blood is not coming to the catheter, the catheterization will be considered unsuccessful. Patients with two unsuccessful attempts per group will be excluded from the study, as more than two unsuccessful attempts may result in infiltration (INS, 2011). Vein visibility after tourniquet application, catheter number used in the procedure, time to determine the appropriate vein, successful catheter placement time, number of attempts for successful catheter placement will be recorded in the intravenous chemotherapy application registration form. The pain and arm comfort levels in the form will be evaluated on a scale ranging from 0 to 10, with 0: none, 10: many, before and after the application (at the 5th, 30th, and 60th minutes).

Implementation of the study in the vascular imaging device group: The patient's vital signs, skin color and skin turgor will be evaluated and recorded in the peripheral intravenous chemotherapy application registration form. After the tourniquet is attached, the stopwatch will be started and the catheter intervention process will be started when the vein visibility reaches the level where the nurse can insert the catheter. The stopwatch will be terminated at the stage of advancing the branule into the vein and fixing it with a plaster. If the catheterization application is successful or unsuccessful in the first attempt, it will be recorded. PIC success will be evaluated according to whether the branule is placed in the vein. Successful catheter insertion will be considered as blood coming into the chamber of the catheter. Patients with two unsuccessful attempts per group will be excluded from the study, as more than two unsuccessful attempts may result in infiltration (INS, 2011). Vein visibility after tourniquet application, catheter number used in the procedure, time to determine the appropriate vein, successful catheter placement time, number of attempts for successful catheter placement will be recorded in the intravenous chemotherapy application registration form. The pain and arm comfort levels in the form will be evaluated on a scale ranging from 0 to 10, with 0: none, 10: many, before and after the application (at the 5th, 30th, and 60th minutes).

Isometric hand exercise: The patients to be included in this group will have applied isometric hand squeeze exercise, which lasted for twenty minutes a day, five days a week, before the PIVK procedure. On the fifth day, the patient's vital signs, skin color and skin turgor will be evaluated and recorded in the peripheral intravenous chemotherapy application registration form. Patients will be told how to use the stress ball 5 minutes before and during the PIVK procedure before the procedure. Patients will be taught to count from one to three and tighten and loosen the stress ball once, and they will be told to continue squeezing and loosening the stress ball in this way until the procedure is over. Focus their attention on the stress ball during the procedure

ELIGIBILITY:
Inclusion Criteria:

* patients who not allergic to any substance,
* patients who not peripheral vascular disease
* patients who not having a chronic disease other than cancer,
* patients who non alcoholic
* patients who non-smoker
* patients who nottaking anticoagulant therapy
* patients who no signs of infiltration and phlebitis, acute trauma around the extremity, inflammation, ecchymosis, hematoma, scar tissue, edema, metal prosthesis, no paralysis,
* patients who no noticeable deformity and thrombocytopenia in the examination,
* patients who no mastectomy was performed,
* patients who do not have communication problems and whose mental level is suitable for participating in the research

Exclusion Criteria:

* patients have advanced reading comprehension problems
* patients have severe hearing impairment
* patients have under 18 years of age,
* patients have who will receive chemotherapy for the first time,
* patients have change chemotherapy cure treatment,
* patients have allergic to any substance,
* patients who did not volunteer to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-05-17 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | through study completion, an average of 1 year
  It is a one-dimensional scale used in the measurement of VAS pain. Among the one-dimensional scales used to determine the severity of pain in patients, it was determined that the VAS measures more sensitively and is more reliable. The scale consists of a 100 mm long horizontal line. On one end are the phrases "No Pain" and on the other end "Unbearable Pain" describing the most severe pain possible. The patient is asked to mark his pain on the scale. The length of the line from the starting point of the scale to the point marked by the patient is measured and recorded in mm.

SECONDARY OUTCOMES:
Arm Comfort Scale | through study completion, an average of 1 year
  The arm comfort has been developed based on VAS. The patient's subjective arm comfort evaluation at the 5th, 30th and 60th minutes before and after the PIVC administeration will be recorded on the form.
  A 10 cm vertical visual analog scale will be used to evaluate the arm comfort felt by individuals during the procedure, with one end showing the discomfort and the other the best possible comfort (Hausfeld et al., 2015).

OTHER OUTCOMES:
Vein Visibility | through study completion, an average of 1 year
  Vein visibility were recorded in real time as excellent = easily visible; medium =moderately visible or only perceived by light touch; poor = not visible and not perceived by touch by the operator student (Aulagnier et al., 2014).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ege, Faculty of Medicine, Hospital of Oncology, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) doesn't share any other researchers. Only research team will see data on IPD. After the data collection phase is completed and turned into a publication, other researchers can access the publication.

REFERENCES:
- [Background] Chiao FB, Resta-Flarer F, Lesser J, Ng J, Ganz A, Pino-Luey D, Bennett H, Perkins C Jr, Witek B. Vein visualization: patient characteristic factors and efficacy of a new infrared vein finder technology. Br J Anaesth. 2013 Jun;110(6):966-71. doi: 10.1093/bja/aet003. Epub 2013 Feb 5. PMID 23384732
- [Background] Chapman LL, Sullivan B, Pacheco AL, Draleau CP, Becker BM. VeinViewer-assisted Intravenous catheter placement in a pediatric emergency department. Acad Emerg Med. 2011 Sep;18(9):966-71. doi: 10.1111/j.1553-2712.2011.01155.x. Epub 2011 Aug 19. PMID 21854488
- [Background] Francisco MD, Chen WF, Pan CT, Lin MC, Wen ZH, Liao CF, Shiue YL. Competitive Real-Time Near Infrared (NIR) Vein Finder Imaging Device to Improve Peripheral Subcutaneous Vein Selection in Venipuncture for Clinical Laboratory Testing. Micromachines (Basel). 2021 Mar 30;12(4):373. doi: 10.3390/mi12040373. PMID 33808493
- [Background] Hausfeld K, Baker RB, Boettcher-Prior P, Hancock D, Helms C, Jablonski T, Lin L, Menne K, Mittermeier J, Morris M. Randomized Prospective Clinical Trial Comparing Room Temperature and Warmed Intravenous Fluid Boluses on Pediatric Patients' Comfort. J Pediatr Nurs. 2015 Nov-Dec;30(6):e3-9. doi: 10.1016/j.pedn.2015.07.006. Epub 2015 Aug 12. PMID 26277355
- [Background] Eren H, Caliskan N. Effect of a Vein Imaging Device and of Fist Clenching on Determination of an Appropriate Vein and on Catheter Placement Time in Patients Receiving Chemotherapy: A Randomized Controlled Trial. Cancer Nurs. 2022 Mar-Apr 01;45(2):105-112. doi: 10.1097/NCC.0000000000000931. PMID 33654007
- [Result] Aulagnier J, Hoc C, Mathieu E, Dreyfus JF, Fischler M, Le Guen M. Efficacy of AccuVein to facilitate peripheral intravenous placement in adults presenting to an emergency department: a randomized clinical trial. Acad Emerg Med. 2014 Aug;21(8):858-63. doi: 10.1111/acem.12437. PMID 25176152